CLINICAL TRIAL: NCT04279340
Title: Correlation Between Chronic Neck Pain and Shoulder Proprioception Among Patient With Cervical Radiculopathy
Brief Title: Correlation Between Chronic Neck Pain and Shoulder Proprioception Among Patients With Cervical Radiculopathy
Status: Completed | Type: Observational
Sponsor: Yasmin Soliman Abdo Soliman (Other)
Responsible Party: Sponsor-Investigator, Yasmin Soliman Abdo Soliman, Correlation between chronic neck pain and shoulder proprioception among patient with cervical radiculopathy., Cairo University
Organization: Cairo University (Other)
Other Study IDs: P.T.REC/012/002255
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Is there correlation between cervical radiculopathy and shoulder proprioception or not?

ELIGIBILITY:
Inclusion Criteria:

* chronic neck pain with unilateral cervical radiculopathy.

Exclusion Criteria:

* has impingement syndrome ,history of instability and any systemic disease.

Ages: 20 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Out patient clinic at faculty of physical therapy
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-07 (Actual)

PRIMARY OUTCOMES:
Shoulder Proprioception among cervical radiculopathy patients | 15 minute
  Percision of repositioning shoulder with closed eyes in patient with chronic neck pain and cervical radiculopathy

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Giza, Egypt